CLINICAL TRIAL: NCT01088074
Title: A Comparative Study of Incision Closure Methods for Total Knee Arthroplasty
Brief Title: A Comparative Study of Incision Closure Methods for Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Southwest Orthopedic Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB1108-0328
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Total Knee Replacement Closure; Wound Closure
Keywords: Total Knee Replacement; Closure Methods
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Histoacryl Tissue Adhesive (Active Comparator): Histoacryl Blue (HAB) Tissue Adhesive (n-butyl-2 cyanoacrylate; B. Braun Corp., Melsungen, Germany). Histocryl is a FDA-approved sterile liquid skin adhesive that has been utilized as a substitute for sutures for wound closure for approximately 40 years.
  Interventions: Device: Histoacryl Tissue Adhesive
- Dermabond (Active Comparator): Dermabond High Viscosity Tissue Adhesive (2-ocytl cyanoacrylate; Ethicon, Somerville, NJ). Dermabond is also a FDA-approved liquid bonding agent that has been utilized for wound closure for approximately 10 years and proven as effective as sutures.
  Interventions: Device: Dermabond
- Staples (Active Comparator): Visistat 35W Stapler (Teleflex Corp, Limerick, PA). The FDA-approved Weck staple system with stainless steel staples has been proven over years of use and remains the standard accepted closure approach due to speed of insertion as well as removal.
  Interventions: Device: Staples
- Running Subcuticular with Monocryl (Active Comparator): Monocryl 4-0 Suture (Ethicon, Somerville, NJ). Monocryl is an FDA-approved absorbable, synthetic, suture indicated for soft tissue approximation.
  Interventions: Device: Monocryl 4-0

INTERVENTIONS:
Device: Histoacryl Tissue Adhesive
  Arms: Histoacryl Tissue Adhesive
Device: Dermabond
  Arms: Dermabond
Device: Staples
  Arms: Staples
Device: Monocryl 4-0
  Arms: Running Subcuticular with Monocryl

SUMMARY:
The aim of the study is to compare incision closure techniques for total knee replacement using a combination of state-of-the-art sutures with tissue adhesives or staples in an effort to identify the best approach with respect to time efficiency, cost, durability, dehiscence, microbial resistance and cosmesis.

The hypothesis is that the combined suture/adhesive approach (sutures for capsule and subcutaneous layers, and tissue adhesive for the final cutaneous layer) or suture/staple approach will be significantly faster and of comparable durability as the conventional exclusive suture approach (sutures used for the capsule, subcutaneous, and cutaneous layers). This is a prospective, randomized, controlled, single site, unblinded (open label) study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included 18 years or older
* TKA scheduled without a bilateral planned within one week of the initial surgery
* Willingness to attend prescribed physical therapy 3 times per week.

Exclusion Criteria:

* Exclusion criteria included medical conditions or personal circumstances that would prevent participation and completion of physical therapy and follow-up visits
* Current participation in another clinical trial
* Preoperative systemic infections
* Uncontrolled diabetes, or diseases or conditions known to effect the wound healing process
* Known hypersensitivity to cyanoacrylate
* Formaldehyde, or the dye D&C Violet #2
* Prior knee hardware fixation devices
* Prior knee incisions greater than 9cm, and arthrofibrosis as evidence by limited ROM less than 80°.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 1/2009-10/2009
  The primary endpoint is the mean procedure time improvement for TKA incision closure using a combined suture/adhesive or suture/staple approach versus suture closure alone.

SECONDARY OUTCOMES:
Mean postop hospital stay | 1/2009-10/2009
  Change in mean postop hospital stay between study and control cohorts

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation for Southwest Orthopedic Research, Houston, Texas, United States